CLINICAL TRIAL: NCT05629286
Title: Immediate Effect of Rigid Taping and Patella Stabilizing Brace on Proprioception, Functionality, and Balance in Patients With Patellofemoral Pain Syndrome
Brief Title: Rigid Taping and Patella Stabilizing Brace Methods in pwPFPS (Patient With Patellofemoral Pain Syndrome)
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: A-9230347
Record Dates: First submitted 2022-11-10; First posted 2022-11-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: McConnell Taping; Patella Stabilazing Brace; Proprioception; Balance; Gait; Functionality
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intervention Group 1: McConnell taping first and then patella stabilizing brace applied to healty participants and patients with PFPS
  Interventions: Device: McConnell taping; Device: Patella Stabilizer Brace
- Intervention Group 2: first patella stabilizing brace and then applied McConnell taping to healty participants and patients with PFPS
  Interventions: Device: McConnell taping; Device: Patella Stabilizer Brace
- No Intervention Group: no intervention to healty participants and patients with PFPS

INTERVENTIONS:
Device: McConnell taping — non-stretch rigid McConnell tape will be applied
  Groups: Intervention Group 1; Intervention Group 2
Device: Patella Stabilizer Brace — An orthotic application that wraps the patellofemoral joint, which has a patellar cavity and supports the patella, and provides stabilization with velcro
  Groups: Intervention Group 1; Intervention Group 2

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common musculoskeletal disease with an annual prevalence of 22.7%. Pain in the anterior of the knee and/or retropatellar and/or peripatellar region patellofemoral compression force increases, squatting, climbing stairs, prolonged sitting is characterized by increased pain related activities such as flexion after.

A large number of different treatment strategies have been proposed to examine these underlying factors and to address the resulting disorders and activity limitations. PFPS in the conservative treatment of patellar taping, stretching the shortened structures, the vastus medialis obliquus, strengthening activity modification, biofeedback, neuromuscular electrical stimulation, ultrasound, and foot orthoses and brace is located. The most frequently used for the treatment of patients with high effect size physiotherapy treatment and exercise training combined treatment in order to control the pain in the short and medium term, while the external knee supports-foot orthoses (brace), kinesiotape, rigid-band is used. It is known that the most commonly recommended external support for patients in the fight against PFPS in the clinical setting is kinesiological taping and brace. However, since kinesiotaping does not show orthotic properties like brace, their comparison with each other and the study of their effects give misleading results. The use of McConnell taping, which can show similar effects with both kinesiotaping and brace, gives clinically positive results. When the literature was examined, there was no study that examined the effectiveness of brace and rigid taping comparatively. In our study, we aim to investigate the extent to which we can change the impaired patella position in PFPS with the use of rigid tape and brace in accordance with this information in the literature and to examine the possible effects of rigid tape and brace, which we will apply to patients with PFPS, on balance, proprioception, gait and functionality in patients. In line with the results we will obtain, it is aimed to increase the effectiveness of treatment and shorten the recovery time by determining the external support that will help patients exercise and their movements in daily life.

H1: McConnell taping and patella stabilizing brace applications applied to patients with PFPS differ from each other in terms of proprioception, functionality, balance and gait parameters.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with PFPS and agreed to voluntary health subjects will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into tree groups. One of the intervention groups will be taped first, then brace; the other will be used brace first, then tape. Healthy individuals will form the control group.

ELIGIBILITY:
Inclusion Criteria:

* being 18-50 years old
* Having been diagnosed with patellofemoral pain syndrome
* BMI <30 kg/m2
* For the last 3 months, the pain in the front of the knee in descending stairs, squatting and functional activities has been > 3 points on the visual analog scale

Exclusion Criteria:

* The presence of an organic lesion (chondromalesia patella, syndrome of excessive lateral pressure, peripatellar bursitis, bening-malignant neoplasm, tendonitis) that can cause pain in the front of the knee
* Having had steroid injections in the knee within the last 6 months and/or having received a physiotherapy program for the knee
* Having undergone lower extremity surgery
* Having a diagnosis of Grade 2 and above osteoarthritis according to Kellgren Lawrence
* Presence of Patellar Tendinopathy
* Presence of a history of trauma to the lower extremities
* The presence of neurological problems that will affect balance and walking
* Having any rheumatological disease
* The use of an assistive device for the ambulance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have been diagnosed with PFPS, healthy people for control group
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Kujala Patellofemoral Scoring | up to three weeks
  It is a tool that allows functional evaluation in knee complaints due to patellofemoral structure.
Visual Analog Scale | up to three weeks
  The maximum pain intensity assessment of the participants during walking, climbing stairs, descending stairs, sitting and squatting activities will be performed using a 10 cm VAS.

SECONDARY OUTCOMES:
10 Stair Up Test | up to three weeks
  Participants will go up and down with both feet 10 times on a hard step 20 centimeters above the ground.
Squat | up to three weeks
  Participants will be asked to squat from their knees to the point where they cannot see their toes. It will be recorded how many seconds the participants did the 5 repetitions.
Joint Position Sense | up to three weeks
  To assess the knee proprioception of the participants, the method of active presence of a passively determined position will be applied. The patient's extremity is brought to a position and she is expected to bring it to the same position.
Single Leg Stance Test | up to three weeks
  Evaluates the standing balance of the participants.
Y Balance Test | up to three weeks
  The Y balance test is a dynamic test performed in a one-legged posture that requires strength, flexibility, core control and proprioception.

CONTACTS AND LOCATIONS:
Overall Officials: Yildiz Analay Akbaba, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Clifford AM, Dillon S, Hartigan K, O'Leary H, Constantinou M. The effects of McConnell patellofemoral joint and tibial internal rotation limitation taping techniques in people with Patellofemoral pain syndrome. Gait Posture. 2020 Oct;82:266-272. doi: 10.1016/j.gaitpost.2020.09.010. Epub 2020 Sep 15. PMID 32987346
- [Background] Saltychev M, Dutton RA, Laimi K, Beaupre GS, Virolainen P, Fredericson M. Effectiveness of conservative treatment for patellofemoral pain syndrome: A systematic review and meta-analysis. J Rehabil Med. 2018 May 8;50(5):393-401. doi: 10.2340/16501977-2295. PMID 29392329
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] van der Heijden RA, Lankhorst NE, van Linschoten R, Bierma-Zeinstra SM, van Middelkoop M. Exercise for treating patellofemoral pain syndrome. Cochrane Database Syst Rev. 2015 Jan 20;1(1):CD010387. doi: 10.1002/14651858.CD010387.pub2. PMID 25603546
- [Background] Kurt EE, Buyukturan O, Erdem HR, Tuncay F, Sezgin H. Short-term effects of kinesio tape on joint position sense, isokinetic measurements, and clinical parameters in patellofemoral pain syndrome. J Phys Ther Sci. 2016 Jul;28(7):2034-40. doi: 10.1589/jpts.28.2034. Epub 2016 Jul 29. PMID 27512259
- [Background] Sisk D, Fredericson M. Taping, Bracing, and Injection Treatment for Patellofemoral Pain and Patellar Tendinopathy. Curr Rev Musculoskelet Med. 2020 Aug;13(4):537-544. doi: 10.1007/s12178-020-09646-8. PMID 32500350
- [Background] Barton CJ, Lack S, Hemmings S, Tufail S, Morrissey D. The 'Best Practice Guide to Conservative Management of Patellofemoral Pain': incorporating level 1 evidence with expert clinical reasoning. Br J Sports Med. 2015 Jul;49(14):923-34. doi: 10.1136/bjsports-2014-093637. Epub 2015 Feb 25. PMID 25716151
- [Background] McConnell J. Management of patellofemoral problems. Man Ther. 1996 Mar;1(2):60-6. doi: 10.1054/math.1996.0251. PMID 11386839
- [Background] Deng F, Adams R, Pranata A, Cui F, Han J. Tibial internal and external rotation taping for improving pain in patients with patellofemoral pain syndrome. J Sci Med Sport. 2022 Aug;25(8):644-648. doi: 10.1016/j.jsams.2022.04.003. Epub 2022 Apr 12. PMID 35484009
- [Background] Kuru T, Dereli EE, Yaliman A. Validity of the Turkish version of the Kujala patellofemoral score in patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2010;44(2):152-6. doi: 10.3944/AOTT.2010.2252. PMID 20676018
- [Background] D'hondt NE, Struijs PA, Kerkhoffs GM, Verheul C, Lysens R, Aufdemkampe G, Van Dijk CN. Orthotic devices for treating patellofemoral pain syndrome. Cochrane Database Syst Rev. 2002;(2):CD002267. doi: 10.1002/14651858.CD002267. PMID 12076444
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407
- [Background] Dobson F, Hinman RS, Hall M, Terwee CB, Roos EM, Bennell KL. Measurement properties of performance-based measures to assess physical function in hip and knee osteoarthritis: a systematic review. Osteoarthritis Cartilage. 2012 Dec;20(12):1548-62. doi: 10.1016/j.joca.2012.08.015. Epub 2012 Aug 31. PMID 22944525
- [Background] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777